CLINICAL TRIAL: NCT05200091
Title: Sensorimotor Integration Underlying Balance Control in Individuals With Incomplete Spinal Cord Injury: Assessing Neural Changes After the Injury and Promoting Recovery Through Specific Training
Brief Title: Sensorimotor Integration Underlying Balance Control in Individuals With Incomplete Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Dorothy Barthélemy, Associate professor and researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRIR 1325-0118
Record Dates: First submitted 2021-09-01; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Spinal Cord Injuries
Keywords: Combined explosive strength and balance training; Balance control; Corticospinal tract; Intracortical mechanisms; Vestibular system
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined explosive strength and specific balance training group (Experimental): This group will be formed with participants with incomplete spinal cord injury. This group will perform 4 weeks of combined explosive strength and specific balance training.
  Interventions: Other: Combined explosive strength and specific balance training group
- Spinal cord injury control group (No Intervention): This group will be formed with participants with incomplete spinal cord injury. They will perform all the evaluation before and after a 4-week period of rest (no training).
- Healthy control group (No Intervention): Healthy participants will be recruited based on the age and sex of the participants with incomplete spinal cord injury to realize clinical and neurophysiological cortical evaluations.

INTERVENTIONS:
Other: Combined explosive strength and specific balance training group — Training will consist to perform one hour of combined ankle explosive strength training and specific balance training using randomized perturbations.
  Explosive strength training: Participants will perform only 2 sets of 3 min (12 contractions for each set) for both lower limbs and both ankle plantar- and dorsiflexion movements.
  Balance specific training: Participants will be standing, secured by an adjusted harness, which do not support the weight but is strictly there to prevent a fall. They will have online visual feedback of their CoP via an avatar on the screen in front of them. Each training session will consist of 10 sequences of 3 min, including the 5 different conditions:
  * Forward tilt of base of support;
  * Backward tilt of base of support;
  * Translation forward;
  * Translation backward;
  * Without moving their feet, participants will have to move their avatar to reach different targets placed around them on the screen, at different distance from the center.
  Arms: Combined explosive strength and specific balance training group

SUMMARY:
The objectives of the study are to evaluate a 4-week mixed training paradigm consisting of explosive strength training and balance perturbation training efficacy on balance control during standing and locomotion, and to understand the mechanisms of neuroplasticity that would improve sensorimotor integration at supraspinal and spinal levels.

DETAILED DESCRIPTION:
After obtaining their consent, participants will undertake evaluations at different times:

1. Assessment 1 week prior to training
2. Training over 4 weeks (nature of the training depends on the group)
3. Assessment 1 week after training
4. Assessment 1 month after training (follow-up)

Each assessment will be divided in 2 sessions and data will be collected over 2 days, at one session per day. Days can be consecutive or non-consecutive but will be within a given week. The assessment consists of:

* Session 1 (S1; duration: 3h) will include presentation of the Study and obtainment of consent, clinical tests, galvanic vestibular stimulation testing, postural reactions and gait assessment.
* Session 2 (S2; duration: 3h) will include muscle strength, short-afference inhibition, paired pulse and trans cranial magnetic stimulation conditioning of H reflex.

After the initial assessment, iSCI participants will be separated in 2 groups and will receive combination of explosive strength and balance training or no intervention. The training will span over 12 sessions (3 times per week for 4 weeks) and each training session will last approximately 1h (including effective training and installation periods).

ELIGIBILITY:
FOR PARTICIPANTS WITH SPINAL CORD INJURY

Inclusion Criteria:

* Have an incomplete lesion of spinal cord
* Level of spinal cord lesion between C5 and T12
* At least, 6 months post-injury
* Be considered as AIS C or D
* Be able to stand without support for 15 seconds
* Be able to provide informed consent in English or in French

Exclusion Criteria:

* To have cognitive deficits
* To have personal or family history of epilepsy
* To have suffered moderate or severe traumatic brain injury
* To have cochlear implant

FOR CONTROL PARTICIPANTS

Exclusion Criteria:

* To have orthopedics problems
* To have cognitive deficits
* To have neurological problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in muscles EMG responses following balance perturbation | Pre-intervention, immediately after and one-month after intervention
  Evaluation of the latency on Soleus and Tibialis anterior muscles EMG following backward and forward perturbations will be done.
Change in center of pressure displacement following balance perturbation using a force platform | Pre-intervention, immediately after and one-month after intervention
  Excursion of centre of pressure will be analyzed following forward and backward perturbation.
Change in ankle muscle strength using force transducer | Pre-intervention, immediately after and one-month after intervention
  Evaluation of isometric dorsi- and planti-flexors muscle strength in Newton will be done using a force transducer attached to the participant's feet.

SECONDARY OUTCOMES:
Change in intracortical mechanisms using transcranial magnetic stimulation (TMS) | Pre-intervention, immediately after and one-month after intervention
  A paired-pulses paradigm (two trans cranial magnetic stimulations at motor cortex level) will be used to evaluate the intracortical mechanisms
Change in the influence of peripheral afferents on cortical output using short-afference inhibition | Pre-intervention, immediately after and one-month after intervention
  A stimulation (using TMS) at motor cortex level will be triggered just after a peripheral electrical stimulation of tibial nerve to evaluate the peripheral afferents on cortical output.
Change in the modulation of the H reflex by the corticospinal tract | Pre-intervention, immediately after and one-month after intervention
  A stimulation (using TMS) at motor cortex level will be triggered just before a tibial nerve stimulation to evaluate the modulation of the H reflex by the corticospinal tract.
Change in EMG responses following vestibular stimulations during quiet standing | Pre-intervention, immediately after and one-month after intervention
  Galvanic vestibular stimulation will be triggered during quiet standing. EMG responses of Soleus and Tibialis Anterior muscles will be analyzed.
Change in the excursion of the center of pressure following vestibular stimulations | Pre-intervention, immediately after and one-month after intervention
  Galvanic vestibular stimulation will be triggered during quiet standing. The displacement of the center of pressure will be analyzed using a force platform.

OTHER OUTCOMES:
MOntreal Cognitive Assessment (MoCA) score | Before enrollment
  The maximal score is 30 and minimal score 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromobility lab, Montreal, Quebec, Canada